CLINICAL TRIAL: NCT01474031
Title: Prospective Study Deltamotion - DAA THA Study
Status: Terminated | Type: Observational
Why Stopped: Main investigator has left the department and therefore the study had ended
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: DePuy International (Industry)
Responsible Party: Sponsor
Other Study IDs: s52629
Record Dates: First submitted 2011-11-07; First posted 2011-11-17 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2011-08

CONDITIONS: Arthrosis
Keywords: total hip arthroplasty; biomechanics; direct anterior approach
MeSH Terms: conditions — Osteoarthritis | interventions — Biomechanical Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 20 DAA subjects: 20 DAA subjects: THA with a Deltamotion articulating surface utilizing the Direct Anterior Approach
  Interventions: Other: Biomechanics
- Control group: healthy volunteers
  Interventions: Other: Biomechanics

INTERVENTIONS:
Other: Biomechanics — * Time interval: pre-op - 3m - 6m - 12m
  * Assessment of all subjects:
    * XR
    * Gait analysis with surface EMG and trunk markers:
      * Unipodal standing: 3 trials Right and 3 trials Left on FP
      * Level walking: 3 trials Right and 3 trials Left on FP
      * Chair rise: 3 trials, both legs on FP
      * Stair ascent: 3 trials Right and 3 trials Left on first FP
      * Stair descent: 3 trials Right and 3 trials Left on first FP
      * Squat: 3 trials, both legs on FP
    * Bipodal squat: 3 trials Right and 3 trials Left on FP
  * Functional scores (HHS, UCLA, HOOS, SF-36)

SUMMARY:
1. Introduction Few gait analytical data are available concerning the Direct Anterior Approach (DAA) in total hip arthroplasty (THA). All the studies have focused on immediate post-operative recovery. These studies have in general some important shortcomings in order to accurately evaluate the biomechanics of the replaced hip joint. None of the published reports have reported on consecutive intervals of pre-op - 6w - 3m - 6m - 12m. This is of interest as we know that recovery with other approaches takes >1 year. It might be that the DAA approach leads to normal gait patterns at 3m or 6m and that these patterns do not differ from the normal pattern or at >1y post-op. None of the reports utilized out-of-plane movements such as coming down or up stairs or squads. Utilizing trunk markers is frequently not done but it is important to evaluate the centre of mass position during gait. Very few studies utilize kinetic data, which are important in order to thoroughly evaluate the biomechanics and loading of the hip. And maybe most importantly, the biomechanical effect of the diameter of the articulating surface on gait parameters following the DAA has never been evaluated.

   One of the most important advantages of the DAA is the muscle sparing aspect and the presumption that the femoral anatomy and biomechanics can be more accurately and precisely restored. If the diameter of the articulating surface has then also been reconstructed to the almost anatomical diameter, we can assume that this should be the most optimal reconstruction of the hip joint currently available. This could lead to early return to normal gait, to optimal joint loading and a minimal amount of stress shielding of the femoral bone.

   The aim of this project is to prospectively analyse the biomechanics of the hip joint of a THA with a Deltamotion articulating surface utilizing the Direct Anterior Approach.
2. Materials and Methods Hypothesis: The temporo-spatial parameters (velocity, cadence, step length, and stride length) and gait kinematic and kinetic data (external hip and knee muscle moments) are not significantly different between the study and control group at the evaluated time intervals indicating normal or near normal gait patterns in the early post-operative recovery phase.

DETAILED DESCRIPTION:
Estimated inclusion time: 1 July 2011 - 31 December 2013 Cohorts: 20 DAA subjects - 20 control subjects

Assessments:

* Time interval: pre-op - 3m - 6m - 12m
* Gait analysis with surface EMG and trunk markers:

  * Unipodal standing: 3 trials Right and 3 trials Left on FP
  * Level walking: 3 trials Right and 3 trials Left on FP
  * Chair rise: 3 trials, both legs on FP
  * Stair ascent: 3 trials Right and 3 trials Left on first FP
  * Stair descent: 3 trials Right and 3 trials Left on first FP
  * Squat: 3 trials, both legs on FP
  * Bipodal squat: 3 trials Right and 3 trials Left on FP
* Functional scores (HHS, UCLA, HOOS, SF-36)

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-75 years
* BMI: < 30kg/m2
* Diagnosis: unilateral primary and secondary osteoarthritis treated with the Deltamotion THA with a Corail stem

Exclusion Criteria:

* Osteoarthritis other joints and low back impairment
* LLD > 5mm

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 DAA subjects
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
biomechanics | 0.5 year
  prospectively analyse the biomechanics of the hip joint of a THA with a Deltamotion articulating surface utilizing the Direct Anterior Approach

SECONDARY OUTCOMES:
bone remodelling | 1 year
  assess the femoral bone remodelling around the fully coated Corail stem over the first year post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Kristoff Corten, Doctor, Principal Investigator — UZ Pellenberg
Locations (1):
- UZ Pellenberg, Leuven, Belgium